CLINICAL TRIAL: NCT03401385
Title: Phase 1, Two-part, Multicenter, Open-label, Multiple Dose, First-in-human Study of DS-1062a in Subjects With Advanced Solid Tumors (TROPION-PanTumor01)
Brief Title: First-in-human Study of DS-1062a for Advanced Solid Tumors (TROPION-PanTumor01)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Collaborators: Daiichi Sankyo (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DS1062-A-J101; 173812 (Registry Identifier: JAPIC CTI)
Record Dates: First submitted 2018-01-09; First posted 2018-01-17 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Hormone Receptor Positive Breast Cancer; Triple Negative Breast Cancer; Non-small Cell Lung Cancer
Keywords: Hormone Receptor Positive Breast Cancer; Triple Negative Breast Cancer; Non-small Cell Lung Cancer; Other solid tumors
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Intervention Model Description: Single group, but in two study parts, therefore two sequential arms are identified
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation - All Participants (Experimental): All participants enrolled in the dose escalation part
  Interventions: Drug: Datopotamab Deruxtecan (Dato-DXd)
- Dose Expansion - All Participants (Experimental): All participants enrolled in the dose expansion part
  Interventions: Drug: Datopotamab Deruxtecan (Dato-DXd); Drug: Steroid Containing Mouthwash; Other: Non-Steroid Containing Mouthwash

INTERVENTIONS:
Drug: Datopotamab Deruxtecan (Dato-DXd) — A total anti-TROP2 antibody and MAAA-1181a
  Other Names: DS1062a; Study treatment
Drug: Steroid Containing Mouthwash — A mouthwash containing a steroid ingredient administered in sub-study
  Arms: Dose Expansion - All Participants
Other: Non-Steroid Containing Mouthwash — A mouthwash containing a non-steroid ingredient administered in sub-study
  Arms: Dose Expansion - All Participants

SUMMARY:
This study is one single group of participants with non-small cell lung cancer (NSCLC) who have not been cured by other treatments. It is the first time the drug has been used in humans. There will be two parts and a sub-study.

The primary purpose of the parts are:

* Dose Escalation: To investigate the safety and tolerability and to determine the maximum tolerated dose (MTD) and the recommended dose for expansion (RDE) of DS-1062a
* Dose Expansion: To investigate the safety and tolerability of DS-1062a in additional solid tumors

This study is expected to last approximately 6 years from the time the first participant is enrolled to the time the last subject is off the study. Study sites are located in both the United States and Japan.

The number of treatment cycles is not fixed in this study. Participants who continue to benefit from the study treatment may continue, unless:

* they withdraw
* their disease gets worse
* they experience unacceptable side effects.

The primary purpose of the sub-study is to compare the effectiveness of steroid versus non-steroid mouthwash as prophylaxis against oral mucositis/stomatitis in participants receiving DS-1062a.

The sub-study is a randomized study that will include approximately 76 participants enrolling into the Dose Expansion part.

DETAILED DESCRIPTION:
The dosage strength will change during the study but all participants will receive the same study drug. So the study is not a true 2-arm study, it is a 2-part study.

In both parts, participants with pathologically documented unresectable advanced NSCLC and triple negative breast cancer (TNBC) who have been refractory to or relapsed from standard treatment or for which no standard treatment is available, will be enrolled. In Dose Expansion, additional indications (hormone receptor [HR]-positive human epidermal growth factor receptor 2 [HER2]-negative breast cancer, HR-positive HER2-low breast cancer, HER2-positive breast cancer, small cell lung cancer [SCLC], endometrial cancer, pancreatic adenocarcinoma, HER2-negative gastric/gastroesophageal junction [GEJ] cancer, esophageal cancer, head and neck squamous cell carcinoma [HNSCC], transitional cell carcinoma of the urothelium, colorectal cancer [CRC], platinum-resistant ovarian cancer, platinum-sensitive ovarian cancer, cervical cancer, and castration-resistant prostate cancer [CRPC]) may be evaluated, if the study treatment demonstrates acceptable safety, tolerability and efficacy in NSCLC participants. After the primary analysis, the main (registered) study will be considered complete, but data will be collected from participants who continue receiving study drug.

In the sub-study, the additional indications listed for Dose Expansion (except for head and neck cancer) may be evaluated.

ELIGIBILITY:
Inclusion Criteria

All Participants:

* Has relapsed or progressed following local standard treatments or for which no standard treatment is available.
* Consents to provide mandatory pre-treatment tumor tissue samples for the measurement of TROP2 and other biomarkers. There is no minimum TROP2 expression level required for inclusion.
* Consents to undergo mandatory on-treatment biopsy if clinically feasible and not contraindicated at the time of on-treatment biopsy, and consents to provide the tumor tissue samples from on-treatment biopsy for the measurement of TROP2 level and other biomarkers.
* Is aged ≥18 years old.
* Has an Eastern Cooperative Oncology Group performance status 0-1.
* Has a left ventricular ejection fraction (LVEF) ≥50% by either an ECHO or MUGA within 28 days before enrollment.
* Has measurable disease based on RECIST version1.1.
* Has adequate bone marrow reserve and organ function within 7 days before Cycle 1, Day 1.
* Has an adequate treatment washout period prior to Cycle 1, Day 1.
* If of reproductive/childbearing potential, agrees to use a highly effective from of contraception or avoid intercourse during and upon completion of the study and for at least 7 months for females and 4 months for males after the last dose of study drug, and agrees not to retrieve, freeze or donate sperm or ova starting at Screening and throughout the study period, and at least 7 months for males and 4 months for males after the final study drug administration.
* After being fully informed about their illness and the investigative nature of the protocol (including foreseeable risks and possible toxicities), is willing and able comply with the protocol and to provide written, ethics committee-approved informed consent form before performance of any study-specific procedures or examinations.
* Has a life expectancy of ≥3 months.
* Has no prior treatment with antibody drug conjugate with deruxtecan (including trastuzumab deruxtecan [T-DXd; DS-8201a], and/or patritumab deruxtecan [HER3-DXd; U3-1402]) and/or ifinatamab deruxtecan [I-DXd; DS-7300]. (Note: Participants in the new HR-positive HER2-low breast cancer cohort is required to have prior treatment with T-DXd and must not have been treated with any other deruxtecan ADC besides T-DXd.)
* Has no prior treatment with trophoblast cell surface antigen 2 (TROP2)-targeted therapy.

Additional Inclusion Criteria for NSCLC participants:

- Has a pathologically documented unresectable advanced NSCLC disease not amenable to curative therapy.

Additional Inclusion Criteria for TNBC participants:

* Has a pathologically documented advanced/unresectable or metastatic breast cancer with HR- (estrogen and progesterone receptor) negative disease and HER2 negative expression according to the American Society of Clinical Oncology - College of American Pathologists guidelines (ASCO-CAP).

Additional Inclusion Criteria for HR positive, HER2-negative participants:

* Pathologically documented unresectable or metastatic breast cancer that is:

  * HER2-negative
  * Positive for estrogen receptor and/or progesterone receptor
  * Is documented refractory or resistant to endocrine therapy
  * Was previously treated with a minimum of 1 and a maximum of 3 prior lines of chemotherapy in the advanced/metastatic setting

Additional Inclusion Criteria for Small-cell lung cancer (SCLC) participants:

* Pathologically documented unresectable or metastatic, and/or extensive-stage SCLC that was previously treated with 1 to 2 prior lines of therapy including platinum-based chemotherapy and immune checkpoint inhibitor.
* No prior exposure to topotecan and/or irinotecan.

Additional Inclusion Criteria for Endometrial cancer participants:

* Pathologically documented recurrent or persistent endometrial cancer that relapsed or progressed after any established and/or curative therapies, including at least 1 systemic therapy.

Additional Inclusion Criteria for Pancreatic adenocarcinoma participants:

* Pathologically documented unresectable or metastatic pancreatic cancer that was previously treated with at least 1 prior line of systemic therapy in neoadjuvant, adjuvant, locally advanced or metastatic setting.

Additional Inclusion Criteria for HER2-negative gastroesophageal cancer participants:

* Pathologically documented unresectable or metastatic adenocarcinoma of the stomach or esophagus, including the gastroesophagel junction (GEJ) that was previously treated with at least 1 prior line of systemic therapy.
* No known history of HER2-positivity (defined as Immunohistochemistry IHC 3+ or IHC 2+ and in situ hybridization ISH+) as classified by ASCO-CAP at any time.

Additional Inclusion Criteria for Esophageal cancer participants:

* Pathologically documented unresectable or metastatic squamous cell carcinoma of the esophagus that was previously treated with at least 1 prior line of therapy including platinum-based chemotherapy.

Additional Inclusion Criteria for Head and neck squamous cell carcinoma (HNSCC) participants:

* Pathologically documented unresectable or metastatic HNSCC that was previously treated with 1-3 prior lines of therapy including platinum and ICI (in combination or sequential), in the advanced or metastatic setting.

Additional Inclusion Criteria for participants with advanced-stage urothelial cancer:

* Pathologically documented unresectable, locally advanced or metastatic, urothelial carcinoma (transitional cell and mixed transitional/non-transitional cell histologies) of the urothelium (including renal pelvis, ureters, urinary bladder, and urethra) that was previously treated with at least 1 prior line of therapy including an ICI.

Additional Inclusion Criteria for Colorectal cancer (CRC) participants:

* Pathologically documented unresectable or metastatic CRC that was previously treated with, or were not considered candidates for, available therapies including fluoropyrimidine-based chemotherapy, an anti-vascular. endothelial growth factor therapy, and an anti-epidermal growth factor (EGFR) therapy.
* Has not progressed or relapsed within 6 months of therapy with irinotecan.

Additional Inclusion Criteria for Platinum-resistant ovarian cancer participants:

* Pathologically documented unresectable or metastatic ovarian cancer that:

  * Is epithelial ovarian (including less-common histologies per National Comprehensive Cancer Network (NCCN).
  * Has relapsed or progressed within 6 months of platinum-based chemotherapy.

Additional Inclusion Criteria for Platinum-sensitive ovarian cancer participants:

* Pathologically documented unresectable or metastatic ovarian cancer that:

  * Is epithelial ovarian (including less-common histologies per NCCN guidelines), fallopian tube, or primary peritoneal presentation.
  * Has relapsed or progressed at least 6 months after the most recent platinum-based chemotherapy.

Additional Inclusion Criteria for Cervical cancer participants:

- Pathologically documented unresectable or metastatic cervical cancer that relapsed or progressed after at least 1 prior line of systemic therapy.

Additional Inclusion Criteria for Castration-resistant prostate cancer participants:

- Pathologically documented unresectable CRPC that:

* Is adenocarcinoma of the prostate without neuroendocrine differentiation or small cell histology.
* Is surgically or medically castrated, with testosterone levels of less than 50 nanograms per deciliter.
* Objective progression as determined by radiographic progression for participants with measurable disease after androgen deprivation.
* Has relapsed or progressed after at least 1 of the following: abiraterone, enzalutamide, apalutamide or darolutamide.
* Has at least 1 documented lesion on either a bone scan or a CT/MRI scan.
* CRPC subjects will be chemotherapy-naïve.

Additional inclusion criteria for HR-positive HER2-low breast cancer subjects previously treated with T-DXd

* Pathologically documented unresectable or metastatic breast cancer that is:

  * HER2-low, defined as IHC 1+ or IHC 2+ / ISH-negative as classified by ASCO-CAP.
  * Positive for estrogen receptor and/or progesterone receptor
* Was previously treated with T-DXd in the advanced or metastatic setting

Additional Inclusion Criteria for Sub-study:

* Is competent and able to comprehend, sign, and date both the main study and the oral mucositis/stomatitis addendum informed consent forms (ICFs) prior to the start of any sub-study procedure or assessment
* Is willing to comply with the procedures of the sub-study, including keeping a daily questionnaire on oral hygiene and oral mucositis/stomatitis-related symptoms

Exclusion Criteria:

* Has a history of malignancy, other than a tumor type specified in the Inclusion Criteria, except (a) adequately resected non-melanoma skin cancer, (b) curatively treated in situ disease, or (c) other solid tumors curatively treated, with no evidence of disease for ≥3 years.
* Uncontrolled or significant cardiac disease including myocardial infarction or uncontrolled/unstable angina within 6 months prior to Cycle 1 Day 1.
* History of congestive heart failure (New York Heart Association classes II-IV) or uncontrolled or significant cardiac arrhythmia, uncontrolled hypertension(resting systolic blood pressure >180 mm Hg or diastolic blood pressure >110 mm Hg).
* Has a mean corrected QT interval (QTcF) prolongation to >470 ms based on of the screening triplicate 12-lead ECGs.
* Has a history of non-infectious interstitial lung disease (ILD)/pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
* Has clinically significant corneal disease.
* Has an uncontrolled infection requiring IV antibiotics, antivirals, or antifungals. Has active human immunodeficiency virus (HIV) infection that is not well controlled. All of the following criteria are required to define an HIV infection that is well controlled: undetectable viral RNA load, CD4+ count >350, no history of AIDS-defining opportunistic infection within the past 12 months, and stable for at least 4 weeks on the same anti-HIV medications. If an HIV infection meets the above criteria, monitoring of viral RNA load and CD4+ count is recommended. Subjects/participants must be tested for HIV during the Screening Period if acceptable by local regulations or an IRB/IEC.
* Has an active or uncontrolled hepatitis B and/or hepatitis C infection.
* Has spinal cord compression or clinically active brain metastases, defined as untreated and symptomatic, or requiring therapy with steroids or anticonvulsants to control associated symptoms. Participants with clinically inactive brain metastases may be included in the study. A minimum of 2 weeks must have elapsed between the end of whole brain radiotherapy and study enrollment. Participants with treated brain metastases that are no longer symptomatic and who require no treatment with steroids may be included in the study if they have recovered from the acute toxic effect of radiotherapy.
* Is lactating or pregnant as confirmed by pregnancy tests performed within 7 days before enrollment.
* Has unresolved toxicities from previous anticancer therapy.
* Has a concomitant medical condition that would increase the risk of toxicity, in the opinion of the Investigator.
* Has a history of severe hypersensitivity reactions to either the drug substances or inactive ingredients of DS-1062a. Has a history of severe hypersensitivity reaction to other monoclonal antibodies.
* Has any other medical conditions, including cardiac disease or psychological disorders, and/or substance abuse that would increase the safety risk to the participant or interfere with participation of the participant or evaluation of the clinical study in the opinion of the Investigator.
* Clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses including, but not limited to, any underlying pulmonary disorder, or any autoimmune, connective tissue or inflammatory disorders with pulmonary involvement, or prior pneumonectomy.
* Has leptomeningeal carcinomatosis.
* Has substance abuse or any other medical conditions such as clinically significant cardiac or psychological conditions, that may, in the opinion of the investigator, interfere with the participant's participation in the clinical study or evaluation of the clinical study results.
* Psychological, social, familial, or geographical factors that would prevent regular follow-up. Adults under guardianship, curatorship, safeguard of justice, or family empowerment measure are not eligible.
* Otherwise considered inappropriate for the study by the investigator.

Additional Exclusion Criteria for Sub-study:

* Has had any prior oral mucositis/stomatitis that did not resolve within 3 months of signing the ICFs
* Requires oral steroid or steroid nasal spray or inhaler for asthma, chronic obstructive pulmonary disease, or any other reason at the time of randomization
* Requires immunosuppressive drugs at the time of randomization
* Has oral inflammation or infections, including candidiasis (thrush) at the time of randomization
* Has a history of severe hypersensitivity reactions or any other contraindication to steroids or other active principles or excipients of the mouthwash

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 890 (Estimated)
Dates: Start 2018-01-31 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose-limiting toxicities | Within 8 cycles (each cycle is 21 days)
  Dose-limiting toxicities are defined as side effects of a drug or other treatment that are serious enough to prevent an increase in dose or level of that treatment.
Number of participants with adverse events (AEs) | When all participants have either discontinued the study or the last participant enrolled in the study has completed at least 6 months of follow up (approximately 4 years)
Number of participants with Grade >/= 2 oral mucositis/stomatitis in Sub-Study | At 8 weeks

SECONDARY OUTCOMES:
Maximum concentration (Cmax) | Within 8 cycles (each cycle is 21 days for Q3W or 14 days for Q2W)
  Categories: DS-1062a, total anti-TROP2 antibody, MAAA-1181a
Time at which Cmax is reached (Tmax) | Within 8 cycles (each cycle is 21 days for Q3W or 14 days for Q2W)
  Categories: DS-1062a, total anti-TROP2 antibody, MAAA-1181a
Area under the drug concentration-time curve (AUC) to the last observable concentration (AUClast) | Within 8 cycles (each cycle is 21 days for Q3W or 14 days for Q2W)
  Categories: DS-1062a, total anti-TROP2 antibody, MAAA-1181a
AUC during the dosing period (AUCtau) | Within 8 cycles (each cycle is 21 days for Q3W or 14 days for Q2W)
  Categories: DS-1062a, total anti-TROP2 antibody, MAAA-1181a
Minimum observed concentration (Ctrough) | Within 8 cycles (each cycle is 21 days for Q3W or 14 days for Q2W)
  Categories: DS-1062a, total anti-TROP2 antibody, MAAA-1181a

CONTACTS AND LOCATIONS:
Overall Officials: Global Team Leader, Study Director — Daiichi Sankyo
Locations (18):
- United States (13):
  - University of California, Los Angeles, Los Angeles, California
  - Johns Hopkins Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Tisch Cancer Institute, Icahn School of Medicine, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Next Oncology, San Antonio, Texas
  - START Oncology, San Antonio, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
- Japan (5):
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - The Cancer Institute Hospital of Japanese Foundation For Cancer Research, Koto-Ku, Tokyo
  - Showa Medical University Hospital, Shinagawa-Ku, Tokyo
  - National Cancer Center Hospital, Chūōku
  - National Cancer Center Hospital East, Kashiwa

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Bardia A, Krop IE, Kogawa T, Juric D, Tolcher AW, Hamilton EP, Mukohara T, Lisberg A, Shimizu T, Spira AI, Tsurutani J, Damodaran S, Papadopoulos KP, Greenberg J, Kobayashi F, Zebger-Gong H, Wong R, Kawasaki Y, Nakamura T, Meric-Bernstam F. Datopotamab Deruxtecan in Advanced or Metastatic HR+/HER2- and Triple-Negative Breast Cancer: Results From the Phase I TROPION-PanTumor01 Study. J Clin Oncol. 2024 Jul 1;42(19):2281-2294. doi: 10.1200/JCO.23.01909. Epub 2024 Apr 23. PMID 38652877
- [Derived] Heist RS, Sands J, Bardia A, Shimizu T, Lisberg A, Krop I, Yamamoto N, Kogawa T, Al-Hashimi S, Fung SSM, Galor A, Pisetzky F, Basak P, Lau C, Meric-Bernstam F. Clinical management, monitoring, and prophylaxis of adverse events of special interest associated with datopotamab deruxtecan. Cancer Treat Rev. 2024 Apr;125:102720. doi: 10.1016/j.ctrv.2024.102720. Epub 2024 Mar 11. PMID 38502995
- [Derived] Shimizu T, Sands J, Yoh K, Spira A, Garon EB, Kitazono S, Johnson ML, Meric-Bernstam F, Tolcher AW, Yamamoto N, Greenberg J, Kawasaki Y, Zebger-Gong H, Kobayashi F, Phillips P, Lisberg AE, Heist RS. First-in-Human, Phase I Dose-Escalation and Dose-Expansion Study of Trophoblast Cell-Surface Antigen 2-Directed Antibody-Drug Conjugate Datopotamab Deruxtecan in Non-Small-Cell Lung Cancer: TROPION-PanTumor01. J Clin Oncol. 2023 Oct 10;41(29):4678-4687. doi: 10.1200/JCO.23.00059. Epub 2023 Jun 16. PMID 37327461